CLINICAL TRIAL: NCT02830204
Title: Surgical Implantation of TRAnscatheter vaLve in Native Mitral Annular Calcification (SITRAL) Study
Acronym: SITRAL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor Research Institute (Other)
Collaborators: Edwards Lifesciences (Industry)
Responsible Party: Principal Investigator, Robert L. Smith, MD Cardiothoracic Surgeon, Baylor Research Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 016-100
Record Dates: First submitted 2016-05-04; First posted 2016-07-12 (Estimated); Results first posted 2025-02-24 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Mitral Annular Calcification
Keywords: mitral valve regurgitation; mitral valve stenosis
MeSH Terms: conditions — Mitral Valve Insufficiency; Mitral Valve Stenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Mitral Valve Replacement (MVR) with Sapien3 (Experimental): subjects with surgical MVR with Sapien3
  Interventions: Device: Mitral Valve Replacement (MVR) with Sapien3

INTERVENTIONS:
Device: Mitral Valve Replacement (MVR) with Sapien3 — subjects with surgical MVR with Sapien3
  Other Names: MVR

SUMMARY:
The purpose of this study is to establish the safety and feasibility of the Edwards SAPIEN 3 valve in subjects with mitral annular calcification (MAC) associated with mitral stenosis (MS) and/or mitral regurgitation who are at high-risk for mitral valve surgery or deemed inoperable due to the extent of calcification.

DETAILED DESCRIPTION:
Technical Success:

Alive, with

* Successful access, delivery and retrieval of the device delivery system, and
* Deployment and correct positioning (including repositioning/recapture if needed) of the single intended device, and
* No need for additional unplanned or emergency surgery or re-intervention related to the device or access procedure

Device Success:

Alive and stroke free, with

* Original intended device in place, and
* No additional surgical or interventional procedures related to access or the device since completion of the original procedure (i.e., exit from the cath lab/Operating Room(OR)), and
* Intended performance of the device:

  * Structural performance: No migration, embolization, detachment, fracture, hemolysis, thrombosis (including reduced leaflet motion) or endocarditis, etc, and
  * Hemodynamic performance: Maintenance of relief of stenosis or insufficiency without producing the opposite (Stenosis = Mitral Valve Area (MVA) < 1.5cm2 and Mitral Valve (MV) gradient > 5mmHg, Insufficiency = Mitral Regurgitation (MR) >1+), and
  * Absence of para-device complications (e.g., Paravalvular Leak (PVL) > mild, need for a Permanent Pacemaker (PPM), erosion, Annular rupture or Aortic Valve (AV) Groove disruption, Left Ventricular Outflow Tract (LVOT) gradient increase > 10mmHg)

Procedural Success:

Device success, and

* No device or procedure related Serious Adverse Events (SAEs) (Life threatening bleed; major vascular or cardiac structural complications requiring unplanned reintervention or surgery; stage 2 or 3 Acute Kidney Injury (includes new dialysis); Myocardial Infarction (MI) or need for percutaneous coronary intervention (PCI)/coronary artery bypass graft (CABG); severe heart failure (HF) or hypotension requiring intravenous (IV) inotrope, ultrafiltration or mechanical circulatory support; prolonged intubation ( > 48 hours)

6.2 Secondary objective(s)

Device Success (at 6 months and 1 year)

* Subject success 1 year

Device Success:

Alive and stroke free, with

* Original intended device in place, and
* No additional surgical or interventional procedures related to access or the device since completion of the original procedure (i.e., exit from the cath lab/Operating Room (OR)), and
* Intended performance of the device:

  * Structural performance: No migration, embolization, detachment, fracture, hemolysis, thrombosis (including reduced leaflet motion) or endocarditis, etc, and
  * Hemodynamic performance: Maintenance of relief of stenosis or insufficiency without producing the opposite (Stenosis = MVA < 1.5cm2 and MV gradient > 5mmHg, Insufficiency = MR >1+), and
  * Absence of para-device complications (e.g., PVL > mild, need for a PPM, erosion, Annular rupture or AV Groove disruption, LVOT gradient increase > 10mmHg)

ELIGIBILITY:
Inclusion Criteria:

* Subject has severe native mitral annular calcification associated with mitral stenosis and/or regurgitation. Qualifying echo must be within 60 days of the date of the procedure.
* Subject has a clinical indication for mitral valve replacement, as demonstrated by reported New York Heart Association (NYHA) Functional Class II or greater.
* The subject is at least 22 years old.
* The Heart Team agrees that the subject is high risk or inoperable for surgical mitral valve repair or replacement (MVR), based on a conclusion that the probability of death or serious, irreversible morbidity exceeds the probability of meaningful improvement. The following concomitant procedures, are allowed: Maze, Tricuspid Valve Procedures (TVP), and Atrial Fibrillation (AF) ablation, coronary artery bypass grafting and septal myectomy.
* The study subject has been informed of the nature of the study, agrees to its provisions and has provided written informed consent as approved by the Institutional Review Board (IRB) of the respective clinical site.
* The study subject agrees to comply with all required post-procedure follow-up visits

Exclusion Criteria:

* Evidence of an acute myocardial infarction (MI) ≤ 30 days before the intended treatment [defined as: Q wave MI, or non-Q wave MI with total creatine kinase (CK) elevation of creatine kinase-myocardial band (CK-MB) ≥ twice normal in the presence of myocardial band (MB) elevation and/or troponin level elevation (WHO definition)].
* Any therapeutic invasive cardiac procedure resulting in a permanent implant that is performed within 30 days of the index procedure (unless part of planned strategy for treatment of concomitant coronary artery disease).
* Leukopenia (white blood cell count < 2000 cell/mL), acute anemia (hemoglobin < 8 g/dL), or thrombocytopenia (platelet count < 50,000 cell/mL).
* Hemodynamic or respiratory instability requiring vasoactive medications, mechanical ventilation at time of procedure.
* Need for emergency surgery for any reason.
* Severe left ventricular dysfunction with Left Ventricular Ejection Fraction (LVEF) < 30%.
* Severe right ventricular dysfunction
* Pregnancy, lactation, or planning to become pregnant
* Echocardiographic evidence of left ventricular mass, thrombus, or concerns of active infective endocarditis.
* Active upper gastrointestinal (GI) bleeding within 3 months prior to procedure without treatment or 30 days prior to procedure with definitive treatment.
* A known contraindication or hypersensitivity to all anticoagulation regimens, or inability to be maintained on oral anticoagulant following the study procedure.
* End stage renal disease requiring dialysis
* Clinically (by neurologist) or neuroimaging confirmed stroke or transient ischemic attack (TIA) within 30 days of the procedure.
* Estimated life expectancy < 12 months

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2016-11-04 (Actual); Primary Completion 2023-01-03 (Actual); Study Completion 2023-11-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Smith, MD, Principal Investigator — Baylor Research Institute
Locations (6):
- United States (6):
  - St. Vincent Heart Center, Indianapolis, Indiana
  - MHRI Maryland, Baltimore, Maryland
  - Lankenau Institute for Medical Research, Wynnewood, Pennsylvania
  - Baylor College of Medicine, Houston, Texas
  - The Heart Hospital Baylor Plano, Plano, Texas
  - University of Virginia, Charlottesville, Virginia

IPD SHARING:
Plan to Share IPD: No
There is currently no plan to share individual participant data

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a prospective, open-label, multicenter study which identified participants from 8 participating institutions, with 6 different study sites enrolling participants into the trial. First participant enrollment took place on 11/04/2016 with the final participant enrolled on 08/05/2022. All participants were followed for 12 months with the final participant visit taking place on 11/29/2023.
Pre-assignment Details: All participants potentially eligible participants are presented via a case review process where experienced study investigators reviewed all the submitted criteria. Upon case review approval the participant can be enrolled in the study. All approved participants receive the Edwards SAPIEN 3 valve placed in the mitral valve position.
Groups:
- Mitral Valve Replacement With SAPEIN3: Subjects with surgical Mitral Valve Replacement with SAPEIN3 using minimally invasive surgical technique.
Period: Overall Study
Arm/Group | Mitral Valve Replacement With SAPEIN3
Started | 25
Discharge Visit | 18
30 Day Visit | 18
6 Month Visit | 16
Completed | 15
Not Completed | 10
Not completed — Death | 9
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Mitral Valve Replacement With SAPEIN3
Number analyzed (Participants) | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 75.6 (7.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 5
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Body mass index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 29.63 (5.7)
New York Heart Association (NYHA) Classification [Mean (Standard Deviation); unit: units on a scale] — NYHA Classification - The Stages of Heart Failure
  Class I - No symptoms and no limitation in ordinary physical activity, e.g. shortness of breath when walking, climbing stairs etc.
  Class II - Mild symptoms (mild shortness of breath and/or angina) and slight limitation during ordinary activity.
  Class III - Marked limitation in activity due to symptoms, even during less-than-ordinary activity, e.g. walking short distances (20 to 100 m).Comfortable only at rest.
  Class IV - Severe limitations. Experiences symptoms even while at rest. Mostly bedbound patients.
  units on a scale | 2.84 (0.69)
Society of Thoracic Surgeons (STS) Risk of Mortality Mitral Valve Repair [Mean (Standard Deviation); unit: Percentage] — The Society of Thoracic Surgeons (STS) has launched its next-generation Short-Term Risk Calculator to assess risk of operative mortality, major morbidity, and complications after most cardiac procedure categories in the Adult Cardiac Surgery Database (ACSD).
  *The number presented represents the percentage risk of mortality, major morbidity and complications operatively for patients undergoing mitral valve repair.*
  Percentage | 4.00 (2.57)
Society of Thoracic Surgeons (STS) Risk of Mortality Mitral Valve Replacement [Mean (Standard Deviation); unit: Percentage] — The Society of Thoracic Surgeons (STS) has launched its next-generation Short-Term Risk Calculator to assess risk of operative mortality, major morbidity, and complications after most cardiac procedure categories in the Adult Cardiac Surgery Database (ACSD)
  *The number presented represents the percentage risk of mortality, major morbidity and complications operatively for patients undergoing mitral valve replacement.*
  Percentage | 6.13 (2.84)
Forced expiratory volume in 1 second (FEV1%) [Mean (Standard Deviation); unit: Percentage] — a measurement of the volume of air exhaled in the first second after a maximal inhalation, expressed as a percentage of the predicted value. Normal value 80-120%.
  Percentage | 63.47 (26.93)
Diffusing Capacity for Carbon Monoxide (DLCO%) [Mean (Standard Deviation); unit: Percentage] — DLCO measures the amount of carbon monoxide (CO) transferred per minute from alveolar gas to red blood cells (RBCs). This test provides critical insights into the lungs' ability to transfer oxygen from inhaled air to the bloodstream.
  Normal DLCO: Between 75% and 140% of the predicted value. Mildly reduced DLCO: 60% to 75% or the lower limit of normal (LLN) predicted value.
  Severely reduced DLCO: Less than 40% of the predicted value
  Percentage | 56.50 (23.30)
Hypertension [Count of Participants; unit: Participants] | 16
Congestive Heart Failure [Count of Participants; unit: Participants] | 12
Hyperlipidemia [Count of Participants; unit: Participants] | 19
Pulmonary Disease [Count of Participants; unit: Participants] | 10
Concomitant Aortic Valvular Disease [Count of Participants; unit: Participants] | 17
Arrythmia [Count of Participants; unit: Participants] | 11
Prior Myocardial Infarction (MI) [Count of Participants; unit: Participants] | 5
Diabetes [Count of Participants; unit: Participants] | 11
Prior Cardiac Intervention [Count of Participants; unit: Participants] | 16

OUTCOME MEASURES:

1. Primary Outcome: Procedural Success
Description: Procedural Success is defined as:
  1. Device success, and
  2. No device or procedure related serious adverse events (SAEs) (Life threatening bleed; major vascular or cardiac structural complications requiring unplanned reintervention or surgery; stage 2 or 3 acute kidney injury (AKI) (includes new dialysis); myocardial infarction (MI) or need for percutaneous coronary intervention (PCI)/coronary artery bypass graft (CABG); severe heart failure (HF) or hypotension requiring intravenous (IV) inotrope, ultrafiltration or mechanical circulatory support; prolonged intubation ( > 48 hours)
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Mitral Valve Replacement With SAPEIN3
Number analyzed (Participants) | 25
Participants
  Met Outcome Measure | 16
  Did Not Meet Outcome Measure | 9

2. Primary Outcome: Technical Success
Description: Technical Success is defined as:
  1. Alive, with
  2. Successful access, delivery and retrieval of the device delivery system, and
  3. Deployment and correct positioning (including repositioning/recapture if needed) of the single intended device, and
  4. No need for additional unplanned or emergency surgery or re-intervention related to the device or access procedure
Time Frame: Procedure Stop Time
Measure: Count of Participants; unit: Participants
Arm/Group | Mitral Valve Replacement With SAPEIN3
Number analyzed (Participants) | 25
Participants
  Met Outcome Measure | 21
  Did Not Meet Outcome Measure | 4

3. Primary Outcome: Device Success
Description: Device Success is defined as:
  1. Alive and stroke free, with
  2. Original intended device in place, and
  3. No additional surgical or interventional procedures related to access or the device since completion of the original procedure (i.e., exit from the cath lab/operating room (OR)), and
  4. Intended performance of the device:
     1. Structural performance: No migration, embolization, detachment, fracture, hemolysis, thrombosis (including reduced leaflet motion) or endocarditis, etc, and
     2. Hemodynamic performance: Maintenance of relief of stenosis or insufficiency without producing the opposite (Stenosis = mitral valve area (MVA) < 1.5cm2 and mitral valve (MV) gradient > 5mmHg, Insufficiency = mitral regurgitation (MR) >1+), and
     3. Absence of para-device complications (e.g., paravalvular leak (PVL) > mild, need for a permanent pacemaker (PPM), erosion, Annular rupture or aortic valve (AV) Groove disruption, left ventricular outflow tract (LVOT) gradient increase > 10mmHg)
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Mitral Valve Replacement With SAPEIN3
Number analyzed (Participants) | 25
Participants
  Known met Outcome Measure | 0
  Unknown | 12
  Did not meet Outcome Measure | 13

4. Secondary Outcome: Device Success
Description: Device Success is defined as:
  1. Alive and stroke free, with
  2. Original intended device in place, and
  3. No additional surgical or interventional procedures related to access or the device since completion of the original procedure (i.e., exit from the cath lab/operating room (OR)), and
  4. Intended performance of the device:
     1. Structural performance: No migration, embolization, detachment, fracture, hemolysis, thrombosis (including reduced leaflet motion) or endocarditis, etc, and
     2. Hemodynamic performance: Maintenance of relief of stenosis or insufficiency without producing the opposite (Stenosis = MVA < 1.5cm2 and MV gradient > 5mmHg, Insufficiency = MR >1+), and
     3. Absence of para-device complications (e.g., PVL > mild, need for a PPM, erosion, Annular rupture or AV Groove disruption, LVOT gradient increase > 10mmHg)
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Mitral Valve Replacement With SAPEIN3
Number analyzed (Participants) | 25
Participants
  Known Met Outcome Measure | 0
  Unknown | 11
  Known Did Not Meet Outcome Measure | 14

5. Secondary Outcome: Device Success
Description: Device Success is defined as:
  1. Alive and stroke free, with
  2. Original intended device in place, and
  3. No additional surgical or interventional procedures related to access or the device since completion of the original procedure (i.e., exit from the cath lab/OR), and
  4. Intended performance of the device:
     1. Structural performance: No migration, embolization, detachment, fracture, hemolysis, thrombosis (including reduced leaflet motion) or endocarditis, etc, and
     2. Hemodynamic performance: Maintenance of relief of stenosis or insufficiency without producing the opposite (Stenosis = MVA < 1.5cm2 and MV gradient > 5mmHg, Insufficiency = MR >1+), and
     3. Absence of para-device complications (e.g., PVL > mild, need for a PPM, erosion, Annular rupture or AV Groove disruption, LVOT gradient increase > 10mmHg)
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Mitral Valve Replacement With SAPEIN3
Number analyzed (Participants) | 25
Participants
  Known Met Outcome Measure | 2
  Unknown | 10
  Known Did Not Meet Outcome Measure | 13

6. Secondary Outcome: Subject Success
Description: Subject Success is defined as:
  All of the following must be present:
  I. Device success (either optimal or acceptable), and II. Patient returned to the pre-procedural setting: and III. No rehospitalizations or reinterventions for the underlying condition (e.g., mitral regurgitation, heart failure); and IV. Improvement from baseline in symptoms (e.g., NYHA improvement by > or = 1 functional class); and V. Improvement from baseline in functional status (e.g., 6-min walk test improvement by > or = 50 m); and VI. Improvement from baseline in quality-of-life (e.g., Kansas City Cardiomyopathy Questionnaire improvement by > or = 10)
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Mitral Valve Replacement With SAPEIN3
Number analyzed (Participants) | 25
Participants
  Known Met Outcome Measure | 0
  Unknown | 10
  Known Did Not Meet Outcome Measure | 15

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Mitral Valve Replacement With SAPEIN3
All-Cause Mortality (participants affected / at risk) | 9/25
Serious Adverse Events (participants affected / at risk) | 20/25
Other Adverse Events (participants affected / at risk) | 24/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Mitral Valve Replacement With SAPEIN3 (N=25)
Bleeding (Surgical and medical procedures) | 3 — Bleeding related to surgical procedure
Arrhythmia and/or Conduction System Injury (Cardiac disorders) | 5
Stroke (Nervous system disorders) | 1
Subarachnoid Hemmorrhage (Nervous system disorders) | 1
Atrioventricular (A-V) Groove Disruption (Cardiac disorders) | 2
Heart Failure (Cardiac disorders) | 2 — New or Worsening Heart Failure
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 3
Hematoma (Blood and lymphatic system disorders) | 2
Pleural Effusion (Cardiac disorders) | 4
Renal Failure or Insufficieny (Renal and urinary disorders) | 3
Left Ventricular Outflow Tract (LVOT) Obstruction (Cardiac disorders) | 1
Hemodynamic Instability (Cardiac disorders) | 1
Kidney Stone (Renal and urinary disorders) | 1
Paravalvular Leak (Cardiac disorders) | 2
Hemolysis (Blood and lymphatic system disorders) | 2
Respirator Failure (Respiratory, thoracic and mediastinal disorders) | 3
Septicemia (Infections and infestations) | 1
Cardiac Arrest (Cardiac disorders) | 2
Acute Cholecystitis (Hepatobiliary disorders) | 1
Multi-System Organ failure (General disorders) | 1
Mitral Stenosis (Cardiac disorders) | 2
Thromboembolism (Blood and lymphatic system disorders) | 1
Right Carotid Injury (Vascular disorders) | 1
Right Ventricular Failure (Cardiac disorders) | 2
Endometrial Cancer (Reproductive system and breast disorders) | 1
Delirium (Psychiatric disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Mitral Valve Replacement With SAPEIN3 (N=25)
Anemia (Blood and lymphatic system disorders) | 8
Bleeding (Surgical and medical procedures) | 4
Arrhythmia and/or Conduction System Injury (Cardiac disorders) | 6
Heart Failure (Cardiac disorders) | 2
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1
Hematoma (Blood and lymphatic system disorders) | 1
Plural Effusion (Cardiac disorders) | 3
Renal Failure or Insufficiency (Renal and urinary disorders) | 4
Vascular Injury (Vascular disorders) | 1
Seroma (Surgical and medical procedures) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 2
Plasma Free Hemoglobin and Haptoglobin Elevated (Blood and lymphatic system disorders) | 3
Troponin Elevated (Cardiac disorders) | 1
Dysphagia (Gastrointestinal disorders) | 1
Alcohol Withdrawal (General disorders) | 1
Chest Pain - non cardiac (General disorders) | 1
Lactate Dehydrogenase (LDH) Elevated (Blood and lymphatic system disorders) | 2
Pulmonary Edema (Respiratory, thoracic and mediastinal disorders) | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2
Edema (Cardiac disorders) | 1
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 1
Prosthetic Valvular Endocarditis (Cardiac disorders) | 1

LIMITATIONS AND CAVEATS:
This study was limited by inadequate data capture and limited availability of full echo results.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2016-02-26): https://cdn.clinicaltrials.gov/large-docs/04/NCT02830204/Prot_SAP_000.pdf
  • Informed Consent Form (2020-10-27): https://cdn.clinicaltrials.gov/large-docs/04/NCT02830204/ICF_001.pdf